CLINICAL TRIAL: NCT04481295
Title: Effect of Pulmonary Rehabilitation Under Different Oxygen Concentration Using High-flow Nasal Cannula
Brief Title: Study on Optimal Oxygen Concentration During Pulmonary Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Hospital Organization Minami Kyoto Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-24
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: High-flow Nasal Cannula; Exercise Capacity; Chronic Respiratory Failure; Optimal SpO2 Value
Keywords: HFNC; 6MWD

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High SpO2 group (Active Comparator): In this group, patients have undergone 4 weeks of pulmonary rehabilitation under the HFNC (FIO2 value that the minimum SpO2 value during pulmonary rehabilitation is 94-96%, and a flow of 10 L/min).
  Interventions: Other: High-flow nasal cannula
- Low SpO2 group (Active Comparator): In this group, patients have undergone 4 weeks of pulmonary rehabilitation under the HFNC (FIO2 value that the minimum SpO2 value during pulmonary rehabilitation is 84-86%, and a flow of 10 L/min).
  Interventions: Other: Low SpO2

INTERVENTIONS:
Other: High-flow nasal cannula — The nasal high flow therapy has enabled high flow oxygen to be derived through nasal cannula. This mode not only allows constant FiO2 during peak inspiratory flow but also confers benefits including a low level of continuous positive airway pressure with increased end-expiratory lung volume and reduced work of breathing, partly through intrinsic positive end-expiration pressure compensation and dead space washout. The inspired gases are warmed and humidified, improving comfort and possibly reducing airway inflammation, leading to improved drainage of respiratory secretions.
  Arms: High SpO2 group
Other: Low SpO2 — Low SpO2
  Arms: Low SpO2 group

SUMMARY:
The purpose of this study is to compare the exercise capacity between high SpO2 (Minimum SpO2 94-96%) value during pulmonary rehabilitation and low SpO2 (Minimum SpO2 84-86%) value during pulmonary rehabilitation for the patients with chronic respiratory failure receiving long-term oxygen therapy.

DETAILED DESCRIPTION:
In patients with chronic respiratory failure, pulmonary rehabilitation is recognized as an evidence-based treatment in improving exercise capacity, muscle strength, dyspnea, and quality of life. However, optimal SpO2 value during pulmonary rehabilitation in patients with chronic respiratory failure receiving long-term oxygen therapy is unclear.

The present study is randomized to compare the effect of exercise capacity between high SpO2 (Minimum SpO2 94-96%) value during pulmonary rehabilitation and low SpO2 (Minimum SpO2 84-86%) value during pulmonary rehabilitation for the patients with chronic respiratory failure receiving long-term oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic respiratory failure receiving long-term oxygen therapy for more than 3 months.

Exclusion Criteria:

* Subjects with severe cardiovascular disease, liver disease, neurological disease, and renal failure.
* Subjects with a history of hospitalization for pneumonia or exacerbation of respiratory failure within the last month.
* Subjects with changes in LTOT prescription flow within the last month
* Subjects who cannot undergo pulmonary rehabilitation due to severe heart failure, arteriosclerosis obliterans or spinal disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-07-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in the six-minutes walking distance prior to and following 4 weeks of pulmonary rehabilitation | four weeks

SECONDARY OUTCOMES:
Change in the six-minutes walking test (lowest SpO2 value etc.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the constant-load exercise test (duration time etc.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the incremental-exercise test (Maximum load value etc.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the body composition measured by InBody (muscle mass et.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the arterial blood gas (PaO2 value etc.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the inflammation marker (CRP etc.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the nutritional status (body mass index(kg/m2) et.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the sympathetic activity (Plasma catecholamine et.) prior to and following 4 weeks of pulmonary rehabilitation | four weeks
Change in the dyspnea (Modified Borg scale) prior to and following 4 weeks of pulmonary rehabilitation | four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: Undecided